CLINICAL TRIAL: NCT02897557
Title: A Prospective Early Feasibility Study to Assess the Performance of the Insulet Artificial Pancreas (AP) System Using the OmniPod® Insulin Management System and the Dexcom G4® Share™ AP System
Brief Title: Insulet Artificial Pancreas Early Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-IDE #1 and 1a
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Cohort in CRC (Experimental): This study is a single-arm, multi-center, observational clinical trial being conducted in a Clinical Research Center (CRC) setting.
  Interventions: Device: Insulet Artificial Pancreas (AP) System

INTERVENTIONS:
Device: Insulet Artificial Pancreas (AP) System

SUMMARY:
The purpose is to perform an early investigation on the safety and performance of an Automated Glucose Control (AGC) algorithm using the OmniPod® Insulin Management System and gather clinical data that will be used to make improvements or modifications to the algorithm for subsequent studies in adults, adolescents and children with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. Age - For the adult cohort: age 18 to 65 years; adolescent cohort: age 12.0 to 17.9 years; pediatric cohort: age 6.0 to 11.9 years
2. Diagnosed with type 1 diabetes for at least 1 year. Diagnosis is based on investigator's clinical judgment.
3. Total daily dose (TDD) of insulin ≥ 0.3 units/kg/day and A1C > 6% at screening
4. Currently using an insulin pump with U-100 rapid-acting insulin analogs and on pump for at least 6 months prior to start of study
5. Willing to use the study CGM device for one week prior to study start and for the duration of the study
6. Willing to use the OmniPod® Insulin Management System during the study
7. Willing to perform all SMBG testing with the study-approved glucose meter at the frequency specified in the study protocol
8. Willing to abide by meal recommendations for breakfast, lunch and dinner during the study
9. Willing to refrain from use of acetaminophen, pseudoephedrine, and supplemental vitamin C (>2000 mg/daily) for the entire duration of participation in the study
10. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent or guardian willing and able to sign the ICF. Subjects aged ≥ 8 years will be asked to sign an assent form.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. A1c >10% at the Screening visit
2. One or more episodes of severe hypoglycemia requiring emergency room (ER) visit or hospitalization within the past 6 months
3. Hypoglycemic unawareness as determined by a score of 4 or more "R" responses on the Clarke Questionnaire
4. One or more episodes of diabetic ketoacidosis requiring ER visit or hospitalization within the past 6 months
5. Used non-insulin anti-diabetic medication within last 30 days
6. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant)
7. Dermatological conditions at the proposed sensor wear sites that in the investigator's opinion could preclude ability to wear the Pod and/or the Dexcom sensor on the abdomen
8. Known history of myocardial infarction (MI) or stroke within the past 6 months
9. Known history of seizure disorder
10. Known history of adrenal insufficiency
11. Current renal or hepatic disease
12. Untreated or unstable hypothyroidism or celiac disease (per investigator's judgment)
13. Currently undergoing cancer treatment
14. Currently undergoing systemic treatment with steroids or immunosuppressive medication
15. History of any chronic infections that would interfere with participation in the study or place study personnel at undue risk due to blood-borne contaminants
16. Current illness that would interfere with participation in the study
17. Untreated or inadequately treated mental illness
18. Current alcohol abuse per investigator's judgment
19. Electrically-powered implants that may be susceptible to RF interference
20. Currently participating in another clinical study testing an investigational drug or device or participation in a clinical study during which an investigational drug was used within the preceding 30 days
21. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic range (defined as <70 mg/dL) | 36 hours
Percentage of time in severe hyperglycemic range (defined as >/=250 mg/dL) | 36 hours

SECONDARY OUTCOMES:
Mean glucose | 36 hours
Percentage of time < 50 mg/dL | 36 hours
Percentage of time < 60 mg/dL | 36 hours
Percentage of time > 180 mg/dL | 36 hours
Percentage of time >/= 300 mg/dL | 36 hours
Percentage of time in the broad euglycemic range (defined as 70-180) mg/dL) | 36 hours
Percentage of time in the tight euglycemic range (defined as 70-140) mg/dL) | 36 hours
Standard deviation and coefficient of variation of CGM values | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - William Sansum Diabetes Center, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado Denver, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No